CLINICAL TRIAL: NCT00436345
Title: A Randomized, Open Label, Multicentre Study to Compare the Pharmaco-economic Implications of an Analgesia Based Regimen With Remifentanil and a Conventional Sedation Based Regimen Using Propofol in Medical and Post-surgical ICU Subjects Requiring Mechanical Ventilation for at Least 2 Days.
Brief Title: Pharmacoeconomic Consequences Of Analgesia in the Intensive Care Unit (ICU)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruitment issues
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108701
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2010-05-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Analgesia
Keywords: analgesia; Mechanical ventilation; pharmaco-economic; ICU
MeSH Terms: conditions — Agnosia | interventions — Remifentanil; Propofol

ARMS (2):
- Remifentanil (Experimental): remifentanil
  Interventions: Drug: Remifentanil
- Propofol (Active Comparator): Propofol infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remifentanil — analgesia in medical and post-surgical Intensive Care Unit subjects requiring mechanical ventilation
  Arms: Remifentanil
Drug: Propofol — conventional sedation in medical and post-surgical Intensive Care Unit subjects requiring mechanical
  Arms: Propofol

SUMMARY:
This study will be a multicentre randomized, open-label, phase IIIb study. This study will evaluate two different techniques of sedation: an analgesia based regimen with remifentanil versus a conventional sedation based regimen using propofol in subjects that require mechanical ventilation for at least 2 days in the ICU. The conventional sedation based regimen will consist of propofol combined with an opioid according to routine clinical practice (morphine, fentanyl, sufentanil or other as required) . The analgesia based regimen will consist of remifentanil, with propofol added on if required.

ELIGIBILITY:
Inclusion Criteria:

* Medical and post-surgical patients admitted to ICU and requiring mechanical ventilation.
* Intubated subjects expected to require mechanical ventilation for longer than 48 hours after starting the study drug.
* Subjects requiring both analgesia and sedation with a regimen comprising a hypnotic agent and an opioid.

Exclusion Criteria:

* Diagnosis: cardiopulmonary resuscitation (CPR) in the previous 24 hours or expecting to require major surgery within the next three days
* Subject who, in the judgement of the investigator, has a life expectancy of 2 days or refrained or refuses full life support, which would limit the care provided
* Concurrent medications:

  * Requires or is likely to require neuromuscular blocking agents by continuous infusion to facilitate mechanical ventilation
  * Has or is likely to receive an epidural block during the treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Italy (6):
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Palermo, Sicily

RESULTS

PARTICIPANT FLOW:
Groups:
- Remifentanil: Infusion started between 6 and 9 ug/kg/h (micrograms per kilogram per hour), and titrated in 1.5 ug/kg/h increments at 5-10 minute intervals to achieve a level of adequate sedation based on investigator clinical judgement. The maximum dose rate was 45 ug/kg/h. Once the remifentanil infusion rate reached 12 ug/kg/h, the sedative infusion (propofol) could be administered if level of sedation was not adequate.
- Propofol: The administration of propofol combined with an opioid (fentanyl, sufentanil, morphine, or other) as required to maintain adequate analgesia/sedation and stable haemodynamics was performed according to routine clinical practice for the investigational site, and in accordance with standard clinical protocols.
Period: Overall Study
Arm/Group | Remifentanil | Propofol
Started | 21 | 18
Completed | 18 | 18
Not Completed | 3 | 0
Not completed — ICU resident beyond follow-up period | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remifentanil | Propofol | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.7) | 60.2 (14.3) | 61.23 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 10 | 11 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 17 | 38
  Asian | 0 | 1 | 1
Simplified acute physiology score (SAPS II) score [Mean (Standard Deviation); unit: Points on a scale] — The SAPS II score consists of adding the points from 17 variables: age, 12 physiological variables, type of admission, and 3 chronic disease variables. These variables are added to give a SAPS II score with a range of 0 ("predicted mortality" 0%) to 163 ("predicted mortality" 100%). SAPS II data were collected from local laboratories for 24 hours following ICU admission.
  Points on a scale | 25.7 (16.7) | 20.9 (16.1) | 23.23 (16.30)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Time on Mechanical Ventilation (Intent-to-Treat Population)
Description: Time from start of mechanical ventilation until actual extubation (the process of removing a tube from the airway).
Time Frame: Up to 38 days (912 hours)
Population: Intent-to-Treat (ITT) Population: all randomised participants who had taken at least one dose of study medication
Measure: Mean (Standard Error); unit: Hours (hr)
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 18
Hours (hr) | 77 (8.31) | 70 (6.48)

2. Secondary Outcome: Duration of Time in Intensive Care Unit (ICU) and Potential Stay in ICU (the Time Expected for Extubation, i.e., the Time Between Intubation and Eligibility for Extubation, According to Investigator's Decision)
Description: Duration of Intensive Care Unit (ICU) stay and the duration of potential stay in the ICU were measured.
Time Frame: Up to 38 days (912 hours)
Population: ITT Population. Only participants with available ICU data were analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 12 | 14
Hours
  Duration of ICU stay | 212.6 (163.4) | 208.5 (185.2)
  Duration of potential ICU stay | 211.3 (161.4) | 208.1 (185.1)

3. Primary Outcome: Duration of Time on Mechanical Ventilation (Modified-Intent-to-Treat Population)
Description: Time from start of mechanical ventilation until actual extubation.
Time Frame: Up to 38 days (912 hours)
Population: Modified-Intent-to-Treat (mITT) Population: all randomised participants who had taken at least one dose of study medication and who had efficacy measurements
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 18
Hours | 77 (8.31) | 70 (6.48)

4. Primary Outcome: Duration of Time on Mechanical Ventilation (Per-Protocol Population)
Description: Time from start of mechanical ventilation until actual extubation
Time Frame: Up to 38 days (912 hours)
Population: Per-Protocol (PP) Population: all participants from the MITT population without any major protocol violation
Measure: Mean (Standard Error); unit: Hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 11 | 13
Hours | 87 (9.47) | 81 (4.71)

5. Secondary Outcome: Duration of Extubation
Description: Duration of extubation was measured.
Time Frame: up to 38 days (912 hours)
Population: ITT Population. Only participants with available extubation data were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 13 | 12
hours | 0.4 (0.5) | 0.7 (0.8)

6. Secondary Outcome: Duration of Weaning
Description: Duration of weaning (the time from the intubation until the recovery of natural respiratory ability) was measured.
Time Frame: up to 38 days (912 hours)
Population: ITT Population. Only participants for which data are available were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 19 | 14
hours | 0.42 (1.0) | 0.26 (0.3)

7. Secondary Outcome: Duration of Remifentanil Infusion (ITT Population)
Description: Data for this measure come from the infusion pump display; the infusion pump infuses medication (analgesics and sedative agents) into the participant's circulatory system.
Time Frame: Up to 10 days (240 hours)
Population: ITT Population. Only participants infused with Remifentanil were analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 0
Hours | 67.7 (60.3) |

8. Secondary Outcome: Duration of Propofol Infusion (ITT Population)
Description: as for outcome 7
Time Frame: up to 10 days (240 hours)
Population: ITT Population. Only participants infused with Propofol were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 13 | 18
hours | 47.6 (41.8) | 86.2 (89.4)

9. Secondary Outcome: Duration of Sufentanil, Fentanil, and Morphine Infusion (ITT Population)
Description: as for outcome 7
Time Frame: up to 10 days (240 hours)
Population: ITT Population. Only participants infused with Sufentanil, Fentanil, and Morphine were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 0 | 8
hours
  Sufentanil, n=8 |  | 51.2 (15.42)
  Fentanil, n=5 |  | 47.5 (40.7)
  Morphine, n=1 |  | 0.03 (0.0)

10. Secondary Outcome: Dose of Remifentanil Administered - Continuous Infusion
Description: Data for this measure come from infusion pump display; the infusion pump infuses medication (analgesics and sedative agents) into the participant's circulatory system.
Time Frame: Up to 10 days
Population: ITT Population. Only participants dosed with Remifentanil were analyzed.
Measure: Mean (Standard Deviation); unit: ug/kg/h (micrograms per kilogram per hr)
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 0
ug/kg/h (micrograms per kilogram per hr) | 10.6 (7.2) |

11. Secondary Outcome: Doses of Sufentanil and Fentanil Administered - Continuous Infusion
Description: as for outcome 10
Time Frame: up to 10 days
Population: ITT Population. Only participants dosed with Remifentanil were analyzed.
Measure: Mean (Standard Deviation); unit: ug/kg/h
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 0 | 8
ug/kg/h
  Sufentanil, n=8 |  | 0.2 (0.1)
  Fentanil, n=5 |  | 5.0 (7.5)

12. Secondary Outcome: Dose of Propofol Administered - Continuous Infusion
Description: as for outcome 10
Time Frame: Up to 10 days
Population: ITT Population. Only participants dosed with Propofol were analyzed.
Measure: Mean (Standard Deviation); unit: mg/kg/h (milligrams per kilogram per hr)
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 13 | 18
mg/kg/h (milligrams per kilogram per hr) | 2.3 (4.0) | 1.8 (1.3)

13. Secondary Outcome: Dose of Morphine Administered - Continuous Infusion
Description: as for outcome 10
Time Frame: up to 10 days
Population: ITT Population. Only participants dosed with Morphine were analyzed.
Measure: Mean (Standard Deviation); unit: mg/kg/h
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 0 | 1
mg/kg/h |  | 4.3 (0.0)

14. Secondary Outcome: Total Dose of Propofol Administered - Bolus
Description: Data from this measure come from infusion pump display; the infusion pump infuses medication (analgesics and sedative agents) into the participant's circulatory system.
Time Frame: Up to 10 days
Population: ITT Population. Only participants dosed with Propofol were analyzed.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 4 | 4
mg/kg | 1.5 (0.4) | 5.5 (4.5)

15. Secondary Outcome: Total Dose of Fentanil Administered - Bolus
Description: as for outcome 10
Time Frame: Up to 10 days
Population: ITT Population. Only participants dosed with Fentanil were analyzed.
Measure: Mean (Standard Deviation); unit: ug/kg
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 0 | 5
ug/kg |  | 5.1 (3.6)

16. Secondary Outcome: Number of Participants Analyzed for Sedation - Agitation Scale (SAS) and Pain Intensity (PI) Scale
Description: Data from participants in the study for which the Sedation-Agitation Scale (SAS) and Pain Intensity (PI) were recorded were analyzed. "Sedation - Agitation" was assessed, using the "Riker Sedation-Agitation Scale" (SAS), by the following 7-point scale: 7, dangerous agitation; 6, very agitated; 5, agitated; 4, calm, cooperative; 3, sedated; 2, very sedated; 1, unarousable. "Pain Intensity" was assessed by the following 6-point Pain Intensity Scale: 1, no pain; 2, mild pain; 3, moderate pain; 4, severe pain; 5 very severe pain; 6, worst possible pain.
Time Frame: Up to 38 Days
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 18
participants
  Screening period | 21 | 18
  Day 1 | 21 | 18
  Day 2 | 18 | 17
  Day 3 | 15 | 14
  Day 4 | 10 | 11
  Day 5 | 6 | 3
  Day 6 | 2 | 2
  Day 7 | 2 | 1
  Day 8 | 1 | 0
  Day 9 | 1 | 0
  Day 10 | 1 | 0
  Extubation period | 12 | 12
  Post-extubation period | 5 | 6

17. Secondary Outcome: Sedation-Agitation From Screening Through the End of Study
Description: "Sedation - Agitation" was assessed, using the "Riker Sedation-Agitation Scale" (SAS), by the following 7-point scale: 7, dangerous agitation; 6, very agitated; 5, agitated; 4, calm, cooperative; 3, sedated; 2, very sedated; 1, unarousable.
Time Frame: Up to 38 days
Population: mITT Population, according to the participants' status
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 18
Points on a scale
  Screening period | 3.5 (1.0) | 3.7 (1.2)
  Day 1 | 3.0 (0.9) | 2.9 (0.8)
  Day 2 | 2.8 (1.0) | 2.9 (0.9)
  Day 3 | 3.1 (0.8) | 3.1 (0.6)
  Day 4 | 3.4 (0.9) | 3.1 (0.6)
  Day 5 | 3.5 (0.4) | 3.1 (1.1)
  Day 6 | 3.9 (0.2) | 2.6 (0.6)
  Extubation period | 3.2 (0.7) | 3.6 (0.4)
  Post-extubation period | 3.8 (0.8) | 4.0 (0.0)

18. Secondary Outcome: Sedation-Agitation for Day 7
Description: as for outcome 17
Time Frame: Day 7
Population: mITT Population according to the participants' status
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 1 | 1
points on a scale | 4.0 (0.0) | 3.3 (0.0)

19. Secondary Outcome: Sedation-Agitation From Day 8 to Day 10
Description: as for outcome 17
Time Frame: Days 8, 9, and 10
Population: mITT Population according to the participants' status
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 1 | 0
points on a scale
  Day 8 | 4.0 (0.0) |
  Day 9 | 3.3 (0.0) |
  Day 10 | 3.6 (0.0) |

20. Secondary Outcome: Number of Participants Analyzed for BIS (Bispectral Index Scale)
Description: Participants in the study for which BIS were evaluated. The BIS monitor provides a single dimensionless number, the BIS value, which ranges from 0 to 100. A BIS value of 0 equals electroencephalogram silence, near 100 is the expected value in a fully awake adult, and between 40 and 60 indicates a level for general anaesthesia.
Time Frame: Up to 38 days
Population: mITT Population
Measure: Number; unit: participants
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 5 | 0
participants
  Screening period | 3 |
  Day 1 | 4 |
  Day 2 | 4 |
  Day 3 | 5 |
  Day 4 | 4 |
  Day 5 | 1 |
  Day 6 | 0 |
  Day 7 | 0 |
  Day 8 | 0 |
  Day 9 | 0 |
  Day 10 | 0 |
  Extubation period | 2 |
  Post-extubation period | 2 |

21. Secondary Outcome: Bispectral Index (BIS)
Description: The BIS monitor provides a single dimensionless number, the BIS value, which ranges from 0 to 100. A BIS value of 0 equals electroencephalogram silence, near 100 is the expected value in a fully awake adult, and between 40 and 60 indicates a level for general anaesthesia.
Time Frame: Screening through End of Study, up to 38 days
Population: mITT Population. Due to the nonmandatory nature of BIS measure in the clinical practice, some participants did not have all the measures for all days in which they were in the study.
Measure: Mean (Standard Deviation); unit: Points on a scale
Groups:
- Remifentanil: Infusion started between 6 and 9 ug/kg/h (micrograms per killograms per hour), and titrated in 1.5 ug/kg/h increments at 5-10 minute intervals to achieve a level of adequate sedation based on investigator clinical judgement. The maximum dose rate was 45ug/kg/h. Once the remifentanil infusion rate reached 12 ug/kg/h, the sedative infusion (propofol) could be administered if level of sedation was not adequate.
Arm/Group | Remifentanil
Number analyzed (Participants) | 5
Points on a scale
  Screening period (n = 3, 0) | 38.0 (4.6)
  Day 1 (n = 4, 0) | 47.3 (18.3)
  Day 2 (n = 4, 0) | 45.6 (16.8)
  Day 3 (n = 5, 0) | 45.8 (17.5)
  Day 4 (n = 4, 0) | 49.7 (13.3)

22. Secondary Outcome: Bispectral Index (BIS) for Day 5
Description: as for outcome 21
Time Frame: Day 5
Population: mITT Population. At Day 5, only one participant remained in the study; the others were already extubated.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 1 | 0
points on a scale | 52.7 (0.0) |

23. Secondary Outcome: Bispectral Index (BIS) for Extubation Period and Post-Extubation Period
Description: as for outcome 21
Time Frame: up to 38 days
Population: mITT Population. The BIS value was recorded only for 2 participants, in the extubation and post-extubation periods.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 2 | 0
points on a scale
  Extubation period | 70.0 (0.0) |
  Post-Extubation period | 71.8 (1.1) |

24. Secondary Outcome: Pain Intensity (PI)
Description: "Pain Intensity" was assessed by the following 6-point Pain Intensity Scale: 1, no pain; 2, mild pain; 3, moderate pain; 4, severe pain; 5 very severe pain; 6, worst possible pain.
Time Frame: Up to 38 days
Population: ITT Population, according to the participants' status. Participants remained in the study until they could be extubated; thus, the number of participants analyzed may vary by day.
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 21 | 18
Points on a scale
  Screening period, n=21, 18 | 1.3 (0.8) | 1.2 (0.5)
  Day 1, n=21, 18 | 1.3 (0.5) | 1.1 (0.2)
  Day 2, n=18, 17 | 1.2 (0.4) | 1.1 (0.2)
  Day 3, n=15, 14 | 1.2 (0.4) | 1.1 (0.3)
  Day 4, n=10, 11 | 1.2 (0.4) | 1.0 (0.1)
  Day 5, n=6, 3 | 1.3 (0.7) | 1.0 (0.0)
  Day 6, n=2, 2 | 1.0 (0.0) | 1.0 (0.0)
  Day 7, n=2, 1 | 1.0 (0.0) | 1.0 (0.0)
  Extubation period, n=12, 12 | 1.4 (0.8) | 1.4 (0.6)
  Post-extubation period, n=5, 6 | 2.0 (1.0) | 1.3 (0.5)

25. Secondary Outcome: Pain Intensity From Day 8 to Day 10
Description: as for outcome 24
Time Frame: Days 8, 9, and 10
Population: mITT Population. Participants remained in the study until they could be extubated; thus, the number of participants analyzed may vary by day.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Remifentanil | Propofol
Number analyzed (Participants) | 1 | 0
points on a scale
  Day 8 | 1.0 (0.0) |
  Day 9 | 1.0 (0.0) |
  Day 10 | 1.0 (0.0) |

ADVERSE EVENTS:
Arm/Group | Remifentanil | Propofol
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/18
Other Adverse Events (participants affected / at risk) | 6 | 3
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Remifentanil | Propofol
Bradycardia (Cardiac disorders) | 0/21 | 1/18
Ascites (Gastrointestinal disorders) | 1/21 | 0/18
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2/21 | 0/18
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1/21 | 0/18
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/21 | 0/18
Hypertension (Vascular disorders) | 5/21 | 1/18
Hypotension (Vascular disorders) | 2/21 | 0/18
Oedema at surgical site (Skin and subcutaneous tissue disorders) | 0/21 | 1/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.